CLINICAL TRIAL: NCT01569178
Title: The Effect of Intracoronary Reinfusion of Bone Marrow-derived Mononuclear Cells(BM-MNC) on All Cause Mortality in Acute Myocardial Infarction.
Brief Title: BAMI. The Effect of Intracoronary Reinfusion of Bone Marrow-derived Mononuclear Cells(BM-MNC) on All Cause Mortality in Acute Myocardial Infarction
Acronym: BAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Anthony Mathur, Clinical Director, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAMI-01
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Infarction; Death
Keywords: stem cells; acute myocardial infarction; heart failure; heart attack; bone marrow; intracoronary reinfusion; bone marrow derived mononuclear cells; Left ventricular function improvement; mortality
MeSH Terms: conditions — Myocardial Infarction; Death; Heart Failure

STUDY DESIGN:
Masking Description: The advanced therapy treatment product used in this trial is open label, hence no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): optimal standard care post myocardial infarction
- Intracoronary Reinfusion of Cells (Experimental): Bone marrow-derived progenitor cells aspiration and Intracoronary reinfusion of the cells
  Interventions: Procedure: Bone Marrow aspiration and intracoronary reinfusion

INTERVENTIONS:
Procedure: Bone Marrow aspiration and intracoronary reinfusion — Bone marrow-derived progenitor cells are obtained from 50ml bone marrow aspirated under local anaesthesia from the iliac crest. Intracoronary infusion of the cells is performed via conventional percutaneous intracoronary intervention techniques using an over-the-wire balloon technique
  Arms: Intracoronary Reinfusion of Cells

SUMMARY:
This is a multinational, multicentre, randomised open-label, controlled, parallel-group phase III study. Its aim is to demonstrate that a single intracoronary infusion of autologous bone marrow-derived mononuclear cells is safe and reduces all-cause mortality in patients with reduced left ventricular ejection fraction(</=45%) after successful reperfusion for acute myocardial infarction when compared to a control group of patients undergoing best medical care.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent form
* men and women of any ethnic origin aged≥18years
* patients with acute ST-elevation myocardial infarction as defined by the universal definition of AMI (including new LBBB)
* Patients with acute ST-elevation myocardial infarction as defined by the universal definition of AMI.
* Successful acute reperfusion therapy (residual stenosis visually <50% and TIMI flow ≥2) within 24 hours of symptom onset or thrombolysis within 12 hours of symptom onset followed by successful percutaneous coronary intervention (PCI) within 24 hours after thrombolysis
* Left ventricular ejection fraction ≤ 45% with significant regional wall motion abnormality assessed by quantitative echocardiography (central, independent core lab analysis) 2 to 6 days after reperfusion therapy
* Open coronary artery suitable for cell infusion supplying the target area of abnormal wall motion

Exclusion Criteria:

* Participation in another clinical trial within 30 days prior randomisation unless non interventional trials or trials where patients are randomised to only standard care and this has been discussed and agreed with the CI/sponsor prior to consenting
* Previously received stem/progenitor cell therapy
* Pregnant or nursing women
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
* Necessity to revascularise additional vessels, outside the target coronary artery at the time of progenitor cell infusion (additional revascularisations after primary PCI and before BM-MNC cell infusion are allowed), unless clinically indicated and according to latest guidelines. This decision should be made at the time of the index procedure and explicitly stated at that time.
* Cardiogenic shock requiring mechanical support
* Platelet count <100.000/µl, or hemoglobin <8.5 g/dl
* Impaired renal function, i.e. creatinine >2.5 mg/dl
* Fever or diarrhoea not responsive to treatment within 4 weeks prior screening
* Cliinically significant bleeding disorder within 3 months prior screening
* Uncontrolled hypertension (systolic >180 mmHg and diastolic >120 mmHg)
* Life expectancy of less than two years from any non-cardiac cause or uncontrolled neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2013-09; Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Time from randomization to all-cause death | for an average of 3 years

SECONDARY OUTCOMES:
Time from randomization to cardiac death | for an average of 3 years
time from randomization to cardiovascular rehospitalisation | for an average of 3 years
  time from randomization to cardiovascular rehospitalisation for recurrent MI, coronary revascularisation procedures, heart failure, Implantation of ICD.CRT device, stroke, syncope or Arrhythmias
incidence and severity of adverse events | for an average of 3 years
bleeding by BARC definition | for an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, MD, FRCP, PhD, Principal Investigator — Queen Mary University of London
Locations (33):
- Belgium (2):
  - Cardiovascular Research Centre VZW, Aalst
  - Katholieke Universiteit Leuven, Leuven
- Fakultni Nemocnice BRNO, Brno, Czechia
- Region Hovedstaden, Copenhagen, Denmark
- Kuopio University Hospital, Kuopio, Finland
- Germany (13):
  - Zentralklinik Bad Berka, Bad Berka
  - Universitätsmedizin Charité Berlin, Berlin
  - UniLinikum Bonn, Bonn
  - Universtitatsklinikum Dusseldorf, Klinik fur Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - HELIOS Klinikum Erfurt GmbH, Erfurt
  - University Hospital Essen, Essen
  - Johann Wolfgang Goethe Universitaet Frankfurt AM MAIN, Frankfurt
  - Klinikum Fulda gAG, Fulda
  - Universitatsmedizin Greifswald Klinik Und Poliklinik Innere Med, Greifswald
  - UKSh Campus Lubeck, Med. Klinik II, Lübeck
  - Krankenhaus Hetzelstift Neustadt, Neustadt
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - University Hospital Ulm, Clinic of Internal Medicine II, Ulm
- Universita Cattolica Del Sacro Cuore, Rome, Italy
- UMC Utrecht, Utrecht, Netherlands
- Spain (10):
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Servico Madrileno De Salud, Madrid
  - Hospital Clinico Salamanca, Salamanca
  - H.U. Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario De Valladolid, Valladolid
  - Hospiatl Universitatio Miguel Servet, Zaragoza
- Cardiocentro Ticino, Lugano, Switzerland
- United Kingdom (2):
  - Queen Mary, University of London (QMUL), London
  - New Cross Hospital, Royal Wolverhampton NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Mathur A, Arnold R, Assmus B, Bartunek J, Belmans A, Bonig H, Crea F, Dimmeler S, Dowlut S, Fernandez-Aviles F, Galinanes M, Garcia-Dorado D, Hartikainen J, Hill J, Hogardt-Noll A, Homsy C, Janssens S, Kala P, Kastrup J, Martin J, Menasche P, Miklik R, Mozid A, San Roman JA, Sanz-Ruiz R, Tendera M, Wojakowski W, Yla-Herttuala S, Zeiher A. The effect of intracoronary infusion of bone marrow-derived mononuclear cells on all-cause mortality in acute myocardial infarction: rationale and design of the BAMI trial. Eur J Heart Fail. 2017 Nov;19(11):1545-1550. doi: 10.1002/ejhf.829. Epub 2017 Sep 25. PMID 28948706